CLINICAL TRIAL: NCT01244438
Title: An Open-Label Phase 2 Pilot Study Evaluating the Activity and Safety of FP 1039 in Subjects With Advanced and/or Recurrent Endometrial Cancers With Specific FGFR2 Mutations
Brief Title: Study of FP-1039 in Subjects With Endometrial Cancers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study FP1039-002 was not feasible. The original assumption was at least 5% of patients screened would qualify, but after screening 70 patients, none qualified.
Sponsor: Five Prime Therapeutics, Inc. (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP1039-002; 2010-024344-15 (EudraCT Number)
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Endometrial Cancers With FGFR2 Mutations
Keywords: endometrial cancer; FGFR2 mutations
MeSH Terms: conditions — Endometrial Neoplasms | interventions — FP-1039

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FP-1039 (Experimental): FP-1039
  Interventions: Drug: FP-1039

INTERVENTIONS:
Drug: FP-1039 — FP-1039 will be administered at a dose up to 16 mg/kg intravenously over 30 minutes once a week.

SUMMARY:
An open-label, non-randomized, single arm study to assess the safety, tolerability, and pharmacokinetics of FP-1039 given by weekly intravenous (IV) administrations in advanced endometrial cancer patients with FGFR2-specific mutations. FP-1039 will be dosed weekly starting at a dose of up to 16 mg/kg.

DETAILED DESCRIPTION:
FP-1039 will be administered intravenously over 30 minutes once a week. All enrolled subjects will be monitored for the occurrence of unacceptable toxicity. Subjects with no evidence of disease progression or unacceptable toxicity after 4 doses of FP-1039 may continue to receive weekly treatment provided there continues to be no evidence of disease progression or unacceptable toxicity. Dosing will be discontinued if a subject has evidence of disease progression. Disease will be assessed approximately every 2 months.

ELIGIBILITY:
Inclusion criteria for study participation:

1. Evidence of histologically or cytologically proven metastatic or locally advanced unresectable endometrial cancer bearing either the S252W or the P243R FGFR2 mutation.
2. Female at least 18 years of age
3. Performance status ≤ 1 on the ECOG Performance Status Scale
4. Adequate cardiac function e.g., NYHA Class I or II
5. Estimated life expectancy of at least 16 weeks
6. Measurable or evaluable disease by physical or radiologic examination
7. Must have recovered from the adverse effects of prior therapy at the time of enrollment to ≤ Grade 1 (excluding alopecia)
8. Meets laboratory criteria as specified per protocol.

Exclusion Criteria for study participation:

1. Prior treatment with an inhibitor of the FGF/FGFR pathway
2. Prior treatment with any of the following:

   * Cytotoxic chemotherapy (including investigational cytotoxic agents) or biologic agents (antibodies, immune modulators, cytokines) within 4 weeks, or nitrosoureas or mitomycin C within 6 weeks prior to the scheduled first dose of FP-1039
   * A small-molecule kinase inhibitor (including investigational small-molecule kinase inhibitors) within 14 days (or 5 half lives of the drug or active metabolites) of the scheduled first dose of FP-1039
   * Any other investigational therapy within 28 days of the first scheduled dose of FP-1039 Note: Any eligibility questions related to prior therapies including the timing from prior therapies should be discussed and a decision agreed on by the Investigator and the Sponsor in writing prior to the subject entering the study
3. Known hypersensitivity to the components of FP-1039
4. Current anticoagulation with therapeutic doses of warfarin (low-dose warfarin ≤ 1mg/day is permitted)
5. PT/INR and/or PTT test results at screening that are above 1.3 x the laboratory ULN.
6. No exclusionary medical history as described per the protocol.
7. Presence of any of the following conditions:

   * Luminal intestinal cancers and/or abdominal carcinomatosis
   * History of abdominal fistula, gastrointestinal perforation, peptic ulcer disease, or intra-abdominal abscess within 6 months prior to study enrollment
   * Other potential risk factors for gastrointestinal perforation (i.e., acute diverticulitis, intra-abdominal abscess, gastrointestinal obstruction)
8. History of organ, bone marrow, or stem cell transplantation
9. Pregnant or breast feeding
10. Clinically apparent CNS metastases or carcinomatous meningitis Note: Subjects with CNS metastases who have completed a course of radiotherapy and who have been on a stable dose of glucocorticoids for at least 4 weeks are eligible.
11. Uncontrolled intercurrent illness including but not limited to an active infection, hypertension, psychiatric, or substance abuse disorders that would preclude consent, limit compliance with study requirements, or confound safety interpretation.
12. Unable or unwilling to abide by the study protocol or cooperate fully with the Investigator or designee

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | up to 1 year
  To assess the response rate of advanced endometrial cancer patients bearing FGFR-specific mutations
Progression-free survival | 6 months
  To assess 6-month progression free survival of advanced endometrial cancer patients bearing FGFR-specific mutations

SECONDARY OUTCOMES:
Safety and tolerability | up to 1 year
  To evaluate the safety and tolerability of FP-1039 in subjects with advanced endometrial cancer
Pharmacokinetics of Plasma | up to 1 year
  To determine pharmacokinetics (PK) plasma concentration at specified times

CONTACTS AND LOCATIONS:
Overall Officials: Harold Keer, MD, PhD, Study Chair — Five Prime Therapeutics, Inc.